CLINICAL TRIAL: NCT04600141
Title: Clinical Efficacy of Heparin and Tocilizumab in Patients With Severe COVID-19 Infection: a Randomized Clinical Trial
Brief Title: Clinical Efficacy of Heparin and Tocilizumab in Patients With Severe COVID-19 Infection
Acronym: HEPMAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar MD, PhD, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPMAB
Record Dates: First submitted 2020-10-22; First posted 2020-10-23 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: COVID-19; Heparin; Tocilizumab
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 - Therapeutic anticoagulation (Active Comparator): * (I) intravenous UFH started at a dose of 18 IU/kg/h, adjusted according to a nomogram to achieve a TTPa of 1.5 to 2.0 times the reference value; OR
  * (II) subcutaneous LMWH - enoxaparin 1 mg / kg per dose every 12 hours.
  Interventions: Drug: Heparin - Therapeutic dosage
- Group 2 - Prophylactic anticoagulation (Active Comparator): * (I) subcutaneous UFH 5,000 IU every 8 hours; OR
  * (II) subcutaneous LMWH - enoxaparin 40 mg daily.
  Interventions: Drug: Heparin - Prophylactic dosage
- Group 3 - Therapeutic anticoagulation with tocilizumab (Experimental): * (I) Intravenous UFH initiated at a dose of 18 IU / kg / h, adjusted according to a nomogram to achieve a TTPa of 1.5 to 2.0 times the reference value associated with 8 mg / kg / tocilizumab infusion / intravenous dose in a single dose; OR
  * Subcutaneous LMWH - enoxaparin 1 mg / kg per dose every 12 hours associated with an infusion of tocilizumab 8 mg / kg / dose in a single dose.
  Interventions: Drug: Tocilizumab; Drug: Heparin - Therapeutic dosage
- Group 4 - Prophylactic anticoagulation with tocilizumab (Experimental): * (I) subcutaneous UFH 5,000 IU every 8 hours associated with an infusion of tocilizumab 8 mg / kg / intravenous dose in a single dose; OR
  * (II) subcutaneous LMWH - enoxaparin 40 mg daily associated with an infusion of tocilizumab 8 mg / kg / intravenous dose in a single dose.
  Interventions: Drug: Tocilizumab; Drug: Heparin - Prophylactic dosage

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab infusion 8mg/kg/dose - Intravenous single dose.
  Arms: Group 3 - Therapeutic anticoagulation with tocilizumab; Group 4 - Prophylactic anticoagulation with tocilizumab
Drug: Heparin - Therapeutic dosage — Intravenous Non-Fractional Heparine (HNF) starting at 18UI/kg/h adjusted according to a nomogram to achieve an Activated Partial Thromboplastin Time (ATTP) from 1.5 To 2.0 times the reference Value; or Low Molecular Weight Heparin (LMWH) subcutaneous dosage of 1mg/kg per dose every 12 hours
  Arms: Group 1 - Therapeutic anticoagulation; Group 3 - Therapeutic anticoagulation with tocilizumab
Drug: Heparin - Prophylactic dosage — Subcutaneous Non-Fractional Heparine 5000U every 8 hours OR Subcutaneous Low Molecular Weight (LMWH) 40mg/day.
  Arms: Group 2 - Prophylactic anticoagulation; Group 4 - Prophylactic anticoagulation with tocilizumab

SUMMARY:
The COVID-19 infection primarily manifests itself as a respiratory tract infection, although new evidence indicates that this disease has systemic involvement involving multiple systems including the cardiovascular, respiratory, gastrointestinal, neurological, hematopoietic and immune systems. Recent studies have shown that in its pathophysiology, inflammation and thrombogenesis predominate, especially in the severe forms of COVID-19. Thus, the investigators hypothesized that the use of heparin and tocilizumab could potencially reduce inflammation and thrombogenesis in patients with severe COVID-19 infection, improving patients outcomes and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Informed consent form signed by the patient or guardian or by audio with the guardian;
* Positive result for COVID-19 in PCR (polymerase chain reaction) in nasopharyngeal swab or tracheal secretion up to 10 days before the inclusion and radiological evidence of COVID-19, by chest radiography or chest computed tomography;
* Need for ≥ 4 L of supplemental oxygen to maintain peripheral oxygen saturation equal to or greater than 93% or need for invasive mechanical ventilation.

Exclusion Criteria:

* Risk of bleeding:

  * Clinical: active bleeding, major surgery in the last 30 days, gastrointestinal bleeding within 30 days;
  * Laboratory: platelet count <50,000, INR> 2 or APTT> 50s;
* Known or suspected adverse reaction to UFH, including heparin-induced thrombocytopenia (TIH);
* Adverse reaction or allergy to tocilizumab;
* Use of any of the following treatments: UFH to treat a thrombotic event within 12 hours before inclusion; HPBM in therapeutic dose within 12 hours before inclusion; warfarin (if used 7 days before and if INR greater than 2; thrombolytic therapy within 3 days before; and use of glycoprotein IIb / IIIa inhibitors within the previous 7 days;
* Pregnant or lactating;
* Absolute indication of anticoagulation due to atrial fibrillation or diagnosed thromboembolic event;
* Refusal by family members and / or patient;
* Active tuberculosis;
* Bacterial infection confirmed by culture;
* Neutropenia (<1000 neutrophils / mm3);
* Use of another immunosuppressive therapy that is not a corticosteroid;
* Septic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with clinical improvement | 30 days
  Proportion of patients with clinical improvement in 30 days, defined by hospital discharge or a reduction of at least 2 points compared to baseline on the ordinal scale recommended by the World Health Organization:
  1. Not hospitalized, with no limitations on activities;
  2. Not hospitalized, but limited to activities;
  3. Hospitalized, with no need for supplemental oxygen;
  4. Hospitalized, needing supplemental oxygen;
  5. Hospitalized, requiring high flow oxygen therapy, non-invasive mechanical ventilation or both;
  6. Hospitalized, requiring ECMO, invasive mechanical ventilation or both;
  7. Death.

SECONDARY OUTCOMES:
Hospital and ICU length of stay; | 30 days
  Number of days in hospital and ICU
Duration of invasive mechanical ventilation | 30 days
  Time requiring invasive mechanical ventilation
Duration of vasopressor use | 30 days
  Time of use of vasopressors
Renal failure by AKIN criteria | 30 days
  Renal failure by AKIN criteria in 30 days
Incidence of cardiovascular complications | 30 days
  Myocardial injury; Acute myocardial infarction; Cardiogenic shock; arrhythmias; Myocarditis; Pericarditis; Ventricular dysfunction.
Incidence of venous thromboembolism | 30 days
  Deep vein thrombosis and pulmonary embolism
Mortality | 30, 60 and 90 days
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Ludhmila A Hajjar, MD, PhD, Principal Investigator — InCor - University of Sao Paulo Medical School
Locations (3):
- Brazil (3):
  - Fundação São Francisco Xavier, Ipatinga, Minas Gerais
  - UNIMED Varginha, Varginha, Minas Gerais
  - Universidade Federal de Sergipe, Aracaju, Sergipe

IPD SHARING:
Plan to Share IPD: No